CLINICAL TRIAL: NCT05020457
Title: A Phase II Clinical Study to Evaluate the Efficacy and Safety of SI-B001 in Combination With Chemotherapy in the Treatment of EGFR WT and ALK WT Recurrent and Metastatic Non-small Cell Lung Cancer
Brief Title: SI-B001 Combined With Chemotherapy in the Treatment of EGFR/ALK WT Recurrent or Metastatic NSCLC.
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan Baili Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SI-B001_201
Record Dates: First submitted 2021-08-22; First posted 2021-08-25 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SI-B001 combined with AP or TP_A (Experimental): SI-B001 combined with Platinum-based chemotherapy(AP or TP). Patients enrolled with EGFRwt/ALKwt NSCLC progressed or were intolerant after first-line treatment with anti-PD-1 /L1 mab alone.
  Interventions: Drug: SI-B001; Drug: AP or TP
- SI-B001 combined with Docetaxel_B (Experimental): Patients with EGFRwt/ALKwt non-small cell lung cancer were included and progressed or were intolerant after first-line treatment with platinum-based two-drug chemotherapy plus anti-PD-1 /L1 mab.
  Interventions: Drug: SI-B001; Drug: Docetaxel
- SI-B001 combined with Docetaxel_C (Experimental): Patients enrolled with EGFRwt/ALKwt NSCLC progressed or were intolerant to treatment with anti-PD-1 /PD-L1 monoclonal antibody after first-line or above chemotherapy.
  Interventions: Drug: SI-B001; Drug: Docetaxel

INTERVENTIONS:
Drug: SI-B001 — SI-B001 is administered by intravenous drip once weekly (QW). 120 min ± 10 min after the first intravenous drip, if the infusion reaction is tolerable during the first dose, the subsequent infusion can be completed within 60-120 min (unless agreed or required by the investigator, the infusion time can be extended), if SI-B001 and chemotherapy are used on the same day, the infusion of chemotherapeutic drugs should be continued after the completion of SI-B001 infusion.
Drug: AP or TP — AP or TP should be administered immediately after SI-B001 is completed. The administration of AP or TP should refer to the drug instructions and standard usage.
  Other Names: AP chemotherapy regimen was pemetrexed combined with cisplatin, and TP chemotherapy regimen was paclitaxel combined with cisplatin.
  Arms: SI-B001 combined with AP or TP_A
Drug: Docetaxel — Docetaxel should be administered immediately after SI-B001 is completed. The administration of Docetaxel should refer to the drug instructions and standard usage.
  Arms: SI-B001 combined with Docetaxel_B; SI-B001 combined with Docetaxel_C

SUMMARY:
This multi-center, open label phase II clinical study is performed in patients with locally advanced or metastatic EGFR wild-type ALK wild-type non-small cell lung cancer progressed on prior anti-PD-1 mab ± platinum-based chemotherapy. This study is investigating the safety and efficacy of SI-B001 at optimal combination dose with chemotherapy in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign informed consent forms and follow program requirements；
2. Male or female;
3. Age: ≥ 18 years;
4. Expected survival time ≥ 3 months;
5. Patients with locally advanced or metastatic EGFR wild-type ALK wild-type lung cancer, disease progression or intolerance after first-line treatment with anti-PD-1/PD-L1 antibody, disease progression or intolerance after first-line treatment with anti-PD-1/PD-L1 antibody and platinum-based chemotherapy, or progression or intolerance after first-line treatment with anti-PD-1/PD-L1 monoclonal antibody;
6. The subject agrees to provide archival tumor tissue samples or fresh tissue samples of the primary tumor or metastases within 6 months; if the subject is unable to provide tumor tissue samples and the subject is unable to provide the gene sequencing report, the subject shall agree to complete the ctDNA EGFR detection during the screening period, and can be assessed by the investigator if other inclusion criteria are met;
7. Must have at least one measurable lesion as defined by RECISTv1.1;
8. Performance status score ECOG0 or 1;
9. Toxicities from prior anticancer therapy have recovered to grade ≤ 2 as defined by NCI-CTCAEv5.0 (except alopecia);
10. No severe cardiac dysfunction, left ventricular score ≥ 50%;
11. The level of organ function must meet the following criteria:

    1. Bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 80 × 109/L, hemoglobin ≥ 90 g/L;
    2. Liver function: TBIL ≤ 1.5ULN (total bilirubin ≤ 3ULN for subjects with Gilbert's syndrome, liver cancer or liver metastases); AST and ALT ≤ 2.5ULN for subjects without liver metastases; AST and ALT ≤ 5.0ULN for subjects with liver metastases;
    3. Renal function: creatinine (Cr) ≤ 1.5ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (according to CockcroftandGault formula).
12. Coagulation function: international normalized ratio (INR) ≤ 1.5 × ULN, and activated partial thromboplastin time (APTT) ≤ 1.5ULN;
13. Urine protein ≤ 2 + (measured by dipstick) or < 1000 mg/24 h (urine);
14. Premenopausal women of childbearing potential must have a negative serum or urine pregnancy test 7 before starting treatment and must be non-lactating; all patients (male or female) should take adequate barrier contraception measures throughout the treatment cycle and 6 months after the end of treatment.

Exclusion Criteria:

1. Patients with past use of docetaxel；
2. Prior to signing the informed consent, the gene sequencing or ctDNA testing report of the previous tissue samples indicated the presence of MET 14 exon jump positive, ROS1 rearrangement positive, BRAF V600E mutation positive, NTRK fusion positive, RET rearrangement positive, HER2 mutation positive, HER2 amplification positive, Patients with KRAS G12C mutation positive；
3. Chemotherapy, biotherapy, immunotherapy, radical radiotherapy, and major surgery were used within 4 weeks before the first administration; palliative radiotherapy, targeted therapy (including small-molecule tyrosine kinase inhibitors) and other antitumor therapy were used within 2 weeks;
4. Screening the history of severe heart disease within the first six months, such as: symptomatic congestive heart failure (CHF) ≥2 (CTCAE v5.0) history, New York Heart Society (NYHA) ≥2 heart failure, acute coronary syndrome, etc.;
5. Prolonged QT interval (QTc > 450 msec in men or 470 msec in women), complete left bundle branch block, and Degree III atrioventricular block;
6. Active autoimmune diseases and inflammatory diseases, such as systemic lupus erythematosus, psoriasis requiring systemic treatment, rheumatoid arthritis, inflammatory bowel disease and Hashimoto's thyroiditis, except for type I diabetes, hypothyroidism controllable by replacement therapy only, skin diseases not requiring systemic treatment (such as vitiligo, psoriasis);
7. Other malignancies diagnosed within 5 years prior to first dose,Exceptions include: radical basal cell carcinoma of the skin, scaly cell carcinoma of the skin, and/or radical resection of carcinoma in situ;
8. Hypertension poorly controlled by two antihypertensive drugs (systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg);
9. Pulmonary disease defined as ≥ grade 3 according to CTCAEv5.0, including resting dyspnea, or requiring continuous oxygen therapy, or patients with a history of interstitial lung disease (ILD);
10. Symptoms of active central nervous system metastases.However, patients with stable parenchymal metastases can be stable, and whether it is stable or not is judged by the investigator;
11. Patients with a history of hypersensitivity to recombinant humanized antibodies or human-mouse chimeric antibodies or hypersensitivity to SI-B001 or any of the excipient components of Osimertinib;
12. History of autologous or allogeneic stem cell transplantation;
13. In previous anthracycline (neo) adjuvant therapy, the cumulative dose of anthracycline was > 360 mg/m2;
14. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBV-DNA copy number > 104) or hepatitis C virus (HCV) infection;
15. Active infection requiring systemic treatment, such as severe pneumonia, bacteremia, sepsis, etc.;
16. Received other unmarketed clinical study drugs or treatments within 4 weeks prior to study participation;
17. Other conditions for trial participation were not considered by the investigator to be appropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to approximately 24 months
  Objective Response Rate
Optimal combination dose (only IIa) | Up to approximately 24 months
  Optimal combination dose of SI-B001 with chemotherapy (only IIa)

SECONDARY OUTCOMES:
OS | Up to approximately 24 months
  Overall Survival
PFS | Up to approximately 24 months
  Progression Free Survival
DCR | Up to approximately 24 months
  Disease Control Rate
DOR | Up to approximately 24 months
  Duration of Response
TEAE | Up to approximately 24 months
  Treatment Emergent Adverse Events
Cmax | Up to approximately 24 months
  Maximum serum concentration
Tmax | Up to approximately 24 months
  Time to maximum serum concentration
Ctrough | Up to approximately 24 months
  Minimum serum concentration
ADA | Up to approximately 24 months
  anti-SI-B001 antibody

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Principal Investigator — Sun Yat-sen University Cancer Center (SYSUCC)
Locations (6):
- China (6):
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Sun Yat-sen University Cancer Center (SYSUCC), Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - TaiZhou Hospital of Zhejiang Province, Taizhou, Zhejiang